CLINICAL TRIAL: NCT06803784
Title: Discovery and Validation of Protein Structural Complexes in Circulating Biofluids As Novel Biomarkers for Early Diagnosis, Prognosis and Therapeutic Management of Patients Affected by Neurodegenerative Disorders
Status: Recruiting | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Collaborators: Università del Piemonte Orientale AOU Maggiore della Carità - Novara (Unknown)
Responsible Party: Principal Investigator, Teresa Esposito, Researcher head of the CNR lab, Neuromed IRCCS
Other Study IDs: PNRR-MCNT2-2023-12377375
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease; Amyotrophic Lateral Sclerosis (ALS); Frontotemporal Dementia (FTD); Alzheimer's Disease (AD)
Keywords: protein structural complexes in Neurodegenerative diseases; circulating biomarkers for neurodegenerative diseases
MeSH Terms: conditions — Parkinson Disease; Amyotrophic Lateral Sclerosis; Frontotemporal Dementia | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. blood samples for purification of DNA, plasma, serum and PBMC
  2. Cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Genetic: whole genome sequencing — Genetic: whole genome sequencing PD Partecipants will be assessed for disease progression: Stadio di Hoehn and Yahr, MDS-UPDRS part III, MOCA test, no motor symptoms, therapy and LID occurrence, Sleep disorders. Partecipants will be subjected to peripheral blood sampling for the purification of DNA, plasma, serum, PBMC and generation of hiPSC. DNA of each partecipants we will analysed by whole genome sequencing by next generation sequencing to identify any variant in candidate PD genes
Genetic: whole exome sequencing — Genetic: whole genome sequencing
  AD Partecipants will be assessed for disease progression:
  * assessment of cognitive disorders (MMSE, MOCA test, clock test);
  * assessment of language disorders;
  * current drug therapy (and possible start date of treatment);
  * date of onset of cognitive disorders;
  * acquisition and assessment of imaging data where present (MRI, CT, PET). DNA of each partecipants we will analysed by whole genome sequencing by next generation sequencing to identify any variant in candidate AD genes
Genetic: whole exome sequencing — Genetic: whole genome sequencing
  ALS/FTD Partecipants will be assessed for disease progression:
  * clinical classification according to El Escorial - revised;
  * assessment of cognitive disorders (and classification according to Strong criteria, 2017);
  * assessment of language disorders;
  * ongoing pharmacological therapy (and possible start date of treatment);
  * date of onset of motor and cognitive disorders;
  * acquisition and assessment of imaging data where present (MRI, CT, PET). DNA of each partecipants we will analysed by whole genome sequencing by next generation sequencing to identify any variant in candidate ALS/FTD genes

SUMMARY:
Neurodegenerative disorders (NDDs), such as Parkinson¿s disease (PD), Alzheimer¿s disease (AD), Frontotemporal dementia (FTD) and Amyotrophic Lateral Sclerosis (ALS) are characterized by aggregation and intracellular accumulation of misfolded proteins, which are believed to play a key role in synaptic dysfunction and neuronal death. Protein structural complexes in biofluids have been proposed to mirror pathological conditions suggesting their use as biomarkers for NDDs characterized by protein aggregation. In this framework, we plan to: i) collect a large cohort of NDD and prodromal patients and healthy subjects using standardized clinical and genetics procedures; ii) apply a novel method based on genomics, proteomics and bioinformatic analysis to map protein complexes in biofluids; iii) identify novel circulating biomarkers and correlate them to genetic profiling and disease endophenotypes, and; iv) validate the biological properties in human brain tissue and dopaminergic cultures.

DETAILED DESCRIPTION:
The project is a multicrentric observational study. Institutions involved are:

OU1 - IRCCS INM Neuromed OU2 -University of Piemonte Orientale The project takes advantage from the availability of a large collection of PD samples from familiar and sporadic cases, recruited at IRCCS Neuromed, for which we already collected and stored clinical information, genetic data as well as DNA, serum, plasma and peripheral blood mononuclear cells (PBMCs) for the entire study cohort. induced pluripotent stem cells (iPSC) are available for 6 PD patients and 5 healthy subjects.

The activities of the Operating Unit (OU1) are:

1. Stratification of NDD patients based on genetics and clinical records;
2. Recruitment of CSF sample of NDD patients;
3. Recruitment, WES and bioinformatic analysis of a selected cohort of NDD relatives (200 samples);
4. Bioinformatic analysis to identify protein structural alterations, candidate genes, genetic profiles and deregulatedpathways (OU1/ OU2);
5. Correlation of circulating complex with PD endophenotypes to identify disease biomarkers (OU1/ OU2);
6. Validation in RBD patients and PD relatives to identify early biomarkers for PD (OU1/ OU2);
7. Validation of the protein complexes in human brain slices and analysis of the biological activity of the most relevant CSF and plasmatic complexes in iPSC-derived mdDA neurons (OU1/ OU2).

The activities of the Operating Unit (OU2) are:

1. CSF and plasma sample collection and storage for patients with NDDs;
2. Stratification of patients based on genetics and clinical records (in collaboration with OU1);
3. Detect alterations in protein complexes in CSF samples (100 samples);
4. Identification and validation of CSF biomarkers for PD (100 samples) (in collaboration with OU1);
5. Validate complex biomarkers using immunochemical or targeted analysis on plasma samples (450 samples);
6. Identify potential drug targetable complexes (in collaboration with OU1);
7. Assess whether proteins with structural changes in the CSF/plasma have those changes in the brain as well;
8. Correlate protein structural information with genetics and clinical data (in collaboration with OU1).

ELIGIBILITY:
* Inclusion Criteria:
* Inclusion criteria for PD patients.

For the IRCCS INM Neuromed, patients will be recruited from those affiliated with the Center for the Study and Treatment of Parkinson's Disease of the Neuromed Institute of Pozzilli. Affected subjects will be selected according to the criteria proposed by Gelb et al in 1999. This is a very pragmatic scheme based on the presence of four cardinal signs, the response to a test administration of Levodopa and the absence of atypical signs:

A) Presence of at least 2 of the 4 cardinal signs (tremor, rigidity, bradykinesia, asymmetric onset) one of which must be tremor or bradykinesia; B) Absence of atypical symptoms such as: i) early postural instability, freezing phenomena, cognitive deterioration, hallucinations, pathological involuntary movements, vertical gaze paralysis; ii) proven causes of secondary parkinsonism (focal lesions, drugs, toxic substances); C) Documented response to the use of L-dopa or dapamine agonists (or lack of an adequate therapeutic attempt with L-dopa or dopamine agonists).

* Inclusion criteria forAD patients. Patients will be selected at the Center for Cognitive Disorders and Dementias (CDCD) SCDU Neurology, AOU Maggiore della Carità, Novara. Patients with AD will be included after diagnosis of probable Alzheimer's disease according to the McKhann criteria (2011) and supported by positive biomarkers for amyloidopathy (PET with amyloid tracer or amyloid cerebrospinal fluid dosage).
* Inclusion criteria for FTD/ALS patients. For UPO, patients will be selected at the tertiary center Amyotrophic Lateral Sclerosis - SCDU Neurology, AOU Maggiore della Carità, Novara. Patients with amyotrophic lateral sclerosis will be included following a diagnosis according to the El Escorial criteria - revised (2015): in this regard, only patients with a definite or probable diagnosis supported by laboratory will be included. For patients with FTD, they will be selected at both centers mentioned above with a diagnosis according to the Rascovsky criteria (2011). In this group, the diagnosis will be supported by negative biomarkers for amyloidopathy (PET with amyloid tracer or amyloid cerebrospinal fluid dosage). For patients with concomitant ALS and FTD, the El Escorial criteria (2015) associated with the Strong criteria (2017) will be used.

Exclusion Criteria:

* PD PATIENTS

  * pre-existing psychiatric pathologies;
  * neurodegenerative neurological diseases such as multiple sclerosis, amyotrophic lateral sclerosis, Alzheimer's, neuromuscular diseases, epilepsy;
  * diagnosis of dementia;
* AD/FTD/ALS PATIENTS

  * pre-existing psychiatric pathologies;
  * previous diagnosis of other neurodegenerative neurological diseases;
  * patients unable to sign informed consent.
* CONTROLS

  * pre-existing psychiatric pathologies;
  * neurodegenerative neurological diseases such as Parkinson's, multiple sclerosis, amyotrophic lateral sclerosis, Alzheimer's, neuromuscular diseases, epilepsy;
  * diagnosis of dementia;
  * depression;
  * prolonged intake of anxiolytic, antidepressant, antipsychotic, sleep-inducing, cognitive stimulant drugs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be performed on a total population of 510 subjects (140 PD, 150 AD/ALS/FTD, 120 controls, 100 relatives of patients carrying mutations), of these, 90 patients with a clinical diagnosis of neurodegenerative disease (40 PD cases, 30 AD cases, 20 ALS/FTD cases) will be recruited in this study. The study also includes the recruitment and analysis of 20 control individuals selected among those who will undergo CSF sampling in a diagnostic regimen for non-inflammatory and non-neurodegenerative diseases. The validation cohort, partially already available at the Clinical Centers involved in the study, is composed of 400 subjects of which: 100 PD patients (UO1), 100 AD/FTD/ALS patients (UO2), 100 healthy family members of NDD patients carrying pathogenic mutations and who have not yet developed the disease (UO1) and 100 control individuals (UO1).
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
motor symptoms of PD patients will be evaluated with Hoehn and Yahr (HY) score | 2 years
  The Hoehn and Yahr Scale will be used to measure how Parkinson's symptoms progress and the level of disability. Itincludes stages 1 through 5: Stage 1. Unilateral involvement only, usually with minimal or no functional impairment; Stage 2 = Bilateral disease, without impairment of balance; Stage 3 = Mild to moderate bilateral disease; some postural instability; physically independent. Stage 4 = Severe disability; still able to walk or stand unassisted. Stage 5 = Wheelchair bound or bedridden unless aided.
motor and non motor symptoms of PD patients will be evaluated with MDS-UPDRS | 2 years
  The MDS-UPDRS has four parts, namely, I: Non-motor Experiences of Daily Living; II: Motor Experiences of DailyLiving; III: Motor Examination; IV: Motor Complications. Twenty questions are completed by the patient/caregiver
clinical evaluation of cognitive impairment of PD, AD, ALS/FTD patients | 2 years
  PD patients will be evaluated with the Montreal Cognitive Assessment (MoCA) test. This is a test used by healthcare providers to evaluate people with memory loss or other symptoms of cognitive decline. The MoCA contains 30 questions and checks different types of cognitive or thinking abilities. These include:orientation, short-term memory/delayed recall, executive function/visuospatial ability, clock-drawing test.- assessment of language disorders.
  ALS/FTD - assessment of cognitive disorders (and classification according to Strong criteria, 2017); - assessment of language disorders.
  AD patients: - assessment of cognitive disorders (MMSE, MOCA test, clock test);
  - assessment of language disorders.
clinical evaluation of ALS/FTD patients | 2 years
  Clinical classification according to El Escorial - revised
identification of variants/mutations | 2 years
  PD patients: the number of multiple rare (Minor allele frequency, MAF<0.01) deleterious (missense, non sense, frameshift and splicing) variants in PD genes will be counted in PD patients and unrelated healthy subjects. Case-control assoiciation study will evaluate the PD risk.
  AD, ALS/FTD: deleterious variants (missense, non sense, frameshift and splicing) in responsible genes will be considered.
Identification of protein complexes in CSF | 2 years
  Protein complexes present in the CSF of PD/AD/FTD/ALS patients and control subjects recruited in the two Clinical Centers participating in the study will be analyzed by size exclusion chromatography (SEC) and by label-free proteomic analysis. The complexes will be separated and fractionated by SEC and identified and quantified by mass spectrometers. Statistical analysis will allow to identify the presence/absence or the different abundance of protein complexes in patients compared to controls and therefore the identification of biomarkers and potential therapeutic targets.
Bioinformatic analysis for the identification of proteins and molecular pathways involved | 2 years
  Through advanced bioinformatics analysis, multivariate statistical analysis techniques and machine learning, proteins and molecular pathways involved in different neurodegenerative diseases and their development will be identified. This will allow us to understand and improve the knowledge of these pathologies and to identify potential therapeutic or diagnostic targets/pathways.
Validation of protein complexes in plasma | 2 years
  The key marker protein complexes identified in Phase 1 will be validated in plasma samples from PD/AD/FTD/ALS patients and control subjects through targeted mass spectrometry analyses and through immunochemical technical analyses such as ELISA, Western blot and immunoassays.
Association analysis with endophenotypes | 2 years
  Correlation analyses will be aimed at evaluating whether the presence of aggregates impacts on the age of onset (AAO), neurological symptoms, non-motor symptoms, as well as the response to L-dopa treatment. In addition, genetic data from PD patients will be integrated with biomolecular data to identify altered molecular pathways. ROC curves will be used to evaluate the diagnostic power of the test.
Analysis of the biological impact of protein complexes identified in CSF on the viability of mdDA dopaminergic neurons obtained from iPSCs of patients and controls | 2 years
  Patient and control iPSC lines will be differentiated into mesodiencephalic dopaminergic neurons using published protocols. Cells will be exposed to protein aggregates purified from patient CSF and the cells' vulnerability to neurodegeneration will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: TERESA ESPOSITO, PhD, Principal Investigator — IRCCS INM Neuromed
Locations (1):
- IRCCS INM Neuromed, Pozzilli, Italy, Italy

IPD SHARING:
Plan to Share IPD: No